CLINICAL TRIAL: NCT03388450
Title: Effect of Enteral Nutrition With Omega-3 Fatty Acid in Critically Ill Septic Patients.
Brief Title: Omega-3 Fatty Acid for Critically Ill Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MenoufiaU2015/1ICU
Record Dates: First submitted 2017-12-24; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 (Active Comparator): Patients received enteral nutrition supplemented with 1000 mg omega-3.
  Interventions: Drug: Omega 3
- Placebo (Placebo Comparator): Patients received enteral nutrition supplemented without 1000 mg omega-3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega 3 — Enteral 1000 mg omega 3 fatty acid.
  Other Names: Omega 3 fatty acid
  Arms: Omega 3
Drug: Placebo — Enteral nutrition without omega 3 fatty acid.
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
Sepsis is the most common reason for intensive care unit (ICU) admission. Sepsis flares up the systemic inflammatory response with its mediators. Sepsis treatment protocols have been established in many centres with immune nutrient as adjuvant treatment. Omega-3 fatty acid and other anti-oxidants formulae have been found to improve sepsis outcome. In most of the studies, immune nutrients were giving parenterally, however, nowadays the preferable route of feeding in critically ill patients is enterally. The present study was done to investigate the effect of enteral Omega-3 fatty acid in septic critically ill patients.

DETAILED DESCRIPTION:
A hundred and ten critically ill septic patients were included in the study. Patients were divided into two groups fifty-five patients each. Group A received enteral nutrition supplemented with Omega-3 fatty acid and group B received enteral nutrition without Omega-3. Demographic data, sepsis characteristics, number of patients required invasive ventilation, ventilation days, ICU sequential organ failure assessment score (SOFA), organ failure free-days, haemodynamic failure free-days, ICU stay, ICU and hospital outcomes were recorded.

ELIGIBILITY:
Inclusion Criteria:

* All septic patients who could receive enteral nutrition were included in the study

Exclusion Criteria:

* Patients with end stage liver or renal disease, haemodynamic instability, immunosuppression, gastrointestinal comorbidity, allergic to omega-3, received omega-3 a week prior to ICU admission, patients who expected to live less than 24 hours, and patients who were mechanically ventilated on ICU admission were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Organs dysfunction free days. | 25 days during ICU stay.
  The number of organs dysfunction free days (haemodynamic failure and respiratory failure free days).